CLINICAL TRIAL: NCT03792139
Title: Effects of CYP3A4 Inhibition by Itraconazole on the Pharmacokinetics of LY3200882 in Healthy Subjects
Brief Title: An Interaction Study of LY3200882 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16616; I8X-MC-JECC (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-01-02; First posted 2019-01-03 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3200882 (Experimental): LY3200882 administered orally.
  Interventions: Drug: LY3200882
- Itraconazole + LY3200882 (Experimental): Itraconazole + LY3200882 administered orally.
  Interventions: Drug: LY3200882; Drug: Itraconazole

INTERVENTIONS:
Drug: LY3200882 — Administered orally.
Drug: Itraconazole — Administered orally.
  Arms: Itraconazole + LY3200882

SUMMARY:
The main purpose of this study is to evaluate the effect of itraconazole on the amount of LY3200882 in the blood stream and how long the body takes to get rid of LY3200882. The safety and tolerability of LY3200882 when given with itraconazole will be evaluated. The study is expected to last up to 19 days from the first dose to follow-up (inclusive). Screening will occur up to 28 days prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or postmenopausal females, as determined by medical history and physical examination

Exclusion Criteria:

* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Have used or intend to use over-the-counter or prescription medication including herbal medications within 14 days prior to dosing and during the study (with the exception of vitamins and occasional acetaminophen or ibuprofen, which will be permitted at the discretion of the investigator). Drugs that are known substrates, inducers, or inhibitors of CYP3A4 are specifically excluded within 30 days of dosing and throughout the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-02-23 (Actual); Study Completion 2019-02-23 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Drug Concentration (Cmax) of LY3200882 | Baseline through 72 hours post-dose
  PK: Cmax of LY3200882
PK: Area Under the Concentration Curve (AUC) of LY3200882 | Baseline through 72 hours post-dose
  PK: AUC of LY3200882

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Inc, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No